CLINICAL TRIAL: NCT06844799
Title: A Randomized, Double-blind, Placebo-controlled, Phase 3 Study to Evaluate Efficacy and Safety of HS-20137, an Anti-IL-23 Monoclonal Antibody, in Participants with Moderate-to-severe Plaque Psoriasis
Brief Title: A Study of HS-20137 in Participants with Moderate-to-severe Plaque Psoriasis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-20137-301
Record Dates: First submitted 2025-02-07; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Moderate-to-severe Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- HS-20137 arm1: HS-20137 200mg injection at week 0, 4, 8 and then every 8 weeks thereafter (Experimental)
  Interventions: Drug: HS-20137
- HS-20137 arm 2:HS-20137 200mg injection at week 0, 4, 8 and then every 12 weeks thereafter (Experimental)
  Interventions: Drug: HS-20137
- Placebo arm 1:Placebo at week 0,4,8, and HS-20137 200mg at week 16,20,24 and every8 week thereafter (Experimental)
  Interventions: Drug: Placebo&HS-20137
- Placebo arm 2:Placebo at week 0,4,8, and HS-20137 200mg at week 16,20,24 and every 12week thereafter (Experimental)
  Interventions: Drug: Placebo&HS-20137

INTERVENTIONS:
Drug: HS-20137 — HS-20137 200mg injection at week 0, 4, 8 and then every 8 or 12 weeks.
  Arms: HS-20137 arm 2:HS-20137 200mg injection at week 0, 4, 8 and then every 12 weeks thereafter; HS-20137 arm1: HS-20137 200mg injection at week 0, 4, 8 and then every 8 weeks thereafter
Drug: Placebo&HS-20137 — Placebo injection at week 0, 4, 8, and then HS-20137 200mg injection at week 16, 20, 24, and every 8 or 12 weeks thereafter
  Arms: Placebo arm 1:Placebo at week 0,4,8, and HS-20137 200mg at week 16,20,24 and every8 week thereafter; Placebo arm 2:Placebo at week 0,4,8, and HS-20137 200mg at week 16,20,24 and every 12week thereafter

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of HS-20137 in the treatment of participants with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
HS-20137 is an antibody targeting IL-23, which were recommended biologic agents for the treatment of patients with moderate-to-severe psoriasis. This is a randomized, double-blinded, placebo-controlled phase 3 study, including a 4 weeks screening period, a 52 weeks double-blinded period (placebo-control period in the first 16 weeks) and a 8 weeks follow-up period (total 60 weeks). The hypothesis is that HS-20137 will be more effective in treatment of psoriasis than placebo and well tolerated. Participants with moderate-to-severe plaque psoriasis will be included in this study and received HS-20137 200mg or placebo in week 0, 4, 8 in placebo-control period and then HS-20137 200mg every 8 or 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 and above, male or female;
2. Diagnosed plaque psoriasis for at least 6 months before randomization, with or without psoriatic arthritis;
3. During screening and randomization, the severity of plaque psoriasis was moderate to severe, and the following conditions should be met: a) BSA≥10%; b) PASI≥12; c) sPGA≥3;
4. Suitable for systemic therapy or phototherapy;
5. Voluntarily participate in the research, have the ability and willingness to complete the research according to the research protocol, and sign the informed consent.

Exclusion Criteria:

1. Previous use of biological agents, or allergic reactions to known drug ingredients, or previous severe food or drug allergies;
2. Confirmation of other types of psoriasis, including but not limited to guttiform psoriasis, pustular psoriasis, erythrodermic psoriasis, drug-induced exacerbation of psoriasis (including beta-blockers, non-steroidal anti-inflammatory drugs, antimalarial drugs, interferon, calcium channel blockers, or lithium induced psoriasis) from the screening period to the time before randomization;
3. Other skin lesions, chronic inflammatory diseases or autoimmune diseases, including but not limited to systemic lupus erythematosus, Sjogren's syndrome, skin sclerosis, etc., assessed by the investigator and other factors that may affect the efficacy evaluation or assessed by other researchers before randomization;
4. Primary treatment failure occurred with previous use of similar investigatory drugs (including marketed ulinumab, gusecciumab, Tiricizumab, Lisenciumab, and IL-23 target investigatory drugs under development) (the minimum treatment standard was not reached 12 weeks after the first treatment);
5. Use of the following drugs before randomization:

   1. Use of topical treatment drugs that affect the evaluation of psoriasis within 2 weeks before randomization;
   2. 4 weeks before randomization, Use of phototherapy, traditional systemic therapy drugs, small molecule targeted drugs that may affect the evaluation of psoriasis;
   3. use of TNF-α biologics within 3 months prior to randomization;
   4. use of other biologics for the treatment of psoriasis within 6 months before randomization; e) Use of oral or topical proprietary Chinese medicinesor other Chinese herbal medicines that affect or may affect the evaluation of psoriasis within 4 weeks prior to randomization;

   f) use of lymphocyte migration regulators or B cell and T cell regulators within 3 months before randomization, or 6 months before screening, (whichever is older) use of B-cell-specific scavenging drugs;
6. A history of chronic recurrent infection, or opportunistic infection in the 6 months prior to screening, or hospitalization for a serious infectious disease or intravenous antibiotic use in the 2 months prior to randomization, with a confirmed or suspected illness in the 1 week prior to randomization. And Other circumstances determined by the investigator to be unsuitable for further study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Psoriasis Area and Severity Index (PASI) Score of 90 Percent or Above | At week 16
  Number of participants achieving greater than or equal to 90 percent improvement in PASI at Week 16. PASI is a widely used tool for the measurement of severity of psoriasis. AND, number of participants achieving a physician global assessment (PGA) (0 [none] to 4 [severe]) of cleared or minimal at Week 16
Physician Global Assessment (PGA) score of 0/1 | At week 16
  number of participants achieving a physician global assessment (PGA) (0 [none] to 4 [severe]) of cleared or minimal at Week 16. The PGA is 5-point scale used in clinical trials of various diseases. In this the physician checks the state of the disease and gives them score from 0 (clear) to 4 (severe)

SECONDARY OUTCOMES:
PASI 90 response rate at other visit time points | up to 60 weeks
PASI scores and changes from baseline at each visit time point | up to 60 weeks
PASI 75 response rate and PASI 100 response rate at each visit time point | up to 60 weeks
sPGA 0/1 response rate at other visit time points | during the study period except 16 weeks
sPGA 0 response rate at each visit time point | up to 60 weeks
BSA scores and changes from baseline at each visit time point | up to 60 weeks
  body surface area(BSA):0 = absence of disease, 1 = very mild disease, 2 = mild disease, 3 = moderate disease, and 4 = severe disease